CLINICAL TRIAL: NCT00561145
Title: Impaired Regulation of Energy Balance in Elderly People and the Underlying Physiological Mechanisms.
Brief Title: Impaired Regulation of Energy Balance in Elderly People (Balance Study)
Acronym: Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Dutch Dairy Organization (NZO) (Other)
Responsible Party: Principal Investigator, Lisette de Groot, Professor, Wageningen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL 17278.081.07
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Anorexia of Ageing
Keywords: Anorexia of ageing; Anorexia of aging; Energy balance; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Young men (Experimental): Energy restriction period
  Interventions: Other: Energy restriction period
- Elderly men (Experimental): Energy restriction period
  Interventions: Other: Energy restriction period

INTERVENTIONS:
Other: Energy restriction period — The experiment can be divided in 3 phases, namely (1) run-in phase, (2) energy restriction phase and (3) ad libitum food intake phase. Thus, for all participants the experiment consists of three subsequent phases.

SUMMARY:
Over the past century life expectancy has risen rapidly. As a result, the proportion of elderly people continues to grow. Elderly people probably have an impaired regulation of energy balance (energy intake versus energy expenditure) whereby the underlying physiological mechanisms are not fully understood.

The first objective of this study is to provide further evidence for an age-related failure to regulate energy balance in elderly. If the hypothesis of impaired regulation of energy balance in elderly is confirmed then the second objective becomes to elucidate the underlying physiological mechanisms of the age-related failure to regulate energy intake in elderly.

ELIGIBILITY:
Inclusion Criteria:

* men
* healthy
* 20-40 and 65-85 years of age
* normal weight
* free-living in Wageningen and surrounding

Exclusion Criteria:

* anemia
* diabetes
* restrained eating
* dementia
* weight changes of > 2 kg during the last 2 months

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, Prof, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Result] Winkels RM, Jolink-Stoppelenburg A, de Graaf K, Siebelink E, Mars M, de Groot L. Energy intake compensation after 3 weeks of restricted energy intake in young and elderly men. J Am Med Dir Assoc. 2011 May;12(4):277-86. doi: 10.1016/j.jamda.2010.08.011. Epub 2010 Oct 20. PMID 21527169
- [Derived] Van Bussel IP, Jolink-Stoppelenburg A, De Groot CP, Muller MR, Afman LA. Differences in genome-wide gene expression response in peripheral blood mononuclear cells between young and old men upon caloric restriction. Genes Nutr. 2016 May 6;11:13. doi: 10.1186/s12263-016-0528-0. eCollection 2016. PMID 27551314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited by publishing advertisements in local newspapers and by sending out general e-mails to an e-mail list of persons who had indicated their interest in participating in studies of our university
Groups:
- Young Men: Young men should be 20-40 years of age. Men will be excluded based on the following exclusion criteria:
  body mass index (BMI in kg/m2) less than 20 or higher than 30, adherence to a weight-reduction or medically prescribed diet, dementia (Mini-Mental State Examination score\21), diabetes, anemia, gastrointestinal disorders, use of drugs known to interfere with energy balance, or a history of medical or surgical events known to affect the study outcome.
- Elderly Men: Elderly men should be 65-85 years of age. Men will be excluded based on the following exclusion criteria:
  body mass index (BMI in kg/m2) less than 20 or higher than 30, adherence to a weight-reduction or medically prescribed diet, dementia (Mini-Mental State Examination score\21), diabetes, anemia, gastrointestinal disorders, use of drugs known to interfere with energy balance, or a history of medical or surgical events known to affect the study outcome.
Period: Overall Study
Arm/Group | Young Men | Elderly Men
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Young Men: Young men: 20-40 years of age
- Elderly Men: Elderly men: 65-85 years of age
- Total: Total of all reporting groups
Arm/Group | Young Men | Elderly Men | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 0 | 15
  >=65 years | 0 | 17 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 (1) [20 to 34] | 68 (1) [64 to 85] | 50 (1) [20 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  Netherlands | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Energy Intake Compensation
Description: To assess energy intake compensation, we will assess average energy intake during the ad libitum food intake phase - which is the period after energy restriction- in young men and compare this to average energy intake in older men.
  Average energy intake is assessed by measuring total megajoule of energy intake during nine days of the ad lib phase, and then divide it by nine (MJ/day)
Time Frame: Average intake of energy during ad lib phase (9 days)
Population: completed (see publication)
Measure: Mean (Standard Deviation); unit: MJ/day
Arm/Group | Young Men | Elderly Men
Number analyzed (Participants) | 15 | 17
MJ/day | 1 (1) | 1 (1)

2. Secondary Outcome: Appetite/Satiety Hormones and Questionnaires
Time Frame: Before and after the energy restriction period.
Reporting Status: Not Posted

3. Secondary Outcome: Gastrointestinal Function
Time Frame: Before and after the energy restriction period
Reporting Status: Not Posted

4. Secondary Outcome: Resting Energy Expenditure, Body Composition and Body Weight
Time Frame: Before and after the energy restriction period
Reporting Status: Not Posted

5. Secondary Outcome: Expression of Genes Involved in Energy Metabolism
Time Frame: Before and after the energy restriction period.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the period of the intervention (from enrollment until the end of the ad libitum phase).
Description: We collected data on adverse events (any undesirable experience occurring to a subject during the study). All adverse events reported spontaneously by the subject or observed by the investigator were recorded.
  Serious adverse events were life-threatening events. The chance of those events were considered to be very very low.
Arm/Group | Young Men | Elderly Men
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No